# INFORMED CONSENT FORM AND

# AUTHORIZATION TO USE AND DISCLOSE PROTECTED HEALTH INFORMATION

Sponsor / Study Title: Biomedical Advanced Research and Development Authority

(BARDA)/ "A Two-Period, Two-Sequence, Two-Treatment,

**Single-Dose Crossover Study of Atropine Sulfate** 

Ophthalmic Solution (1%) Administered Sublingually Versus Atropine Sulfate Administered Intramuscularly for

**Bioequivalence Determination Sublingual Atropine Bioequivalence by Route of Administration (SABER)**"

Protocol Number: BP-C-24-0001

**Principal Investigator:** 

(Study Doctor)

Carlos A. Fierro, M.D.

Telephone: (913) 825-4400 (24 Hours)

Address: Johnson County Clin-Trials

16400 College Blvd Lenexa, KS 66219

#### **KEY INFORMATION**

You may be eligible to take part in this research study. This form gives you important information about the study. It describes the purpose of the study, and the risks and possible benefits of participating in this study. Please take enough time to review this information carefully. After you have finished, you should talk to the study doctors and nurses about the study and ask them any questions you may have. You may also wish to talk to others (for example, your friends, family, or other doctors) about your participation in this study. In the end, if you decide to take part in the study, you will be asked to sign this form. Before you sign this form, be sure to understand what the study is about, including the risks and possible benefits to you. Your participation in this study is voluntary, it means that you can choose whether to participate or not.

This research is a Bioequivalence – Bioavailability and pharmacokinetics (PK) study, meaning that this study is comparing how different forms of atropine sulfate (the study drug), specifically atropine sulfate eye drops delivered under the tongue (sublingually) and atropine sulfate injection form delivered using a needle into a muscle of your leg (intramuscular or IM), are similar by measuring the level of study drug that becomes completely available in the bloodstream; also, how the body processes and eliminates the study drug. The goal of this research is to find out if

atropine sulfate eye drops placed under the tongue has a similar effectiveness in the body as the injected form of atropine given IM. There is no direct benefit to you from your participation in this study. Information learned from this study may help other people in the future.

If you choose to participate in this study, you will have 3 in-clinic study visits (Screening Visit, Visit 1, and Visit 2) and one telephone call over a period of approximately 15 days. A Screening Visit will determine if you are eligible to participate in the study. This visit will occur in a single day and last approximately 2-4 hours. At the Screening Visit, if eligible, you will be provided with instructions on how the study visits will be conducted and how you will need to prepare for each visit. You will be asked to return for Visit 1 within the next 3 to 14 days. This visit will last approximately 10 hours. After confirming your eligibility, you will receive a dose of atropine sulfate under the tongue and one dose of atropine sulfate injected into your leg, with the two dosing days being separated by a gap of 5 to 7 days. The order in which the two different dosages will be given to you will be randomly assigned (the same as if you were to flip a coin) at your first visit (Visit 1/Day 1 – or first day of study participation during which you will receive a dose of the study drug). During the study visits when you will receive a dose of study drug either under your tongue or as an injection into your leg, a variety of procedures will be performed including physical examination, blood collections, and a urine test for your use of recreational drugs. You will be asked about your medical history and use of recreational drugs.

After completion of all the requirements at Visit 1, you will be released from the clinic and will be asked to return to the clinic in about 5-7 days for Visit 2. The time between the two clinic visits is called a "washout period". This is necessary to allow your body to remove all traces of atropine from the previous dose so we can compare how your body processes the dose you received by the injection into your leg versus the dose you received under your tongue.

Visit 2 will be like Visit 1. The difference between the two visits will be how atropine will be given to you (under your tongue or by an IM injection into a muscle of your leg). The atropine dose at Visit 2 will be by whatever route you were *not* given during Visit 1. You will also have one follow-up telephone call about 7 days after Visit 2. During this call, the study staff will ask you about any new symptoms and will tell you when you may restart any restricted medications that were withheld during the study period.

You must know the risks and side effects of atropine sulfate and the study procedures. The main risks you should be aware of are a fast heart rate, temporary blurry vision, dry mouth, and a temporary feeling of warmth. A complete list of known risks is provided later in this form.

If you choose to take part in this study and are eligible, you will be expected to attend all study visits and follow instructions for all study procedures.

#### 1. INTRODUCTION

You are deciding if you would like to volunteer for a medical research study. This form will give you more information about the study. Carefully read this form and if you agree to participate in this study, you will have to sign this form. Please ask all the questions you may have before you

decide to participate in the study. Do not sign this form if you have any questions that have not been answered to your full satisfaction and understanding.

The doctor who is conducting this study is being paid by the Sponsor (the Agency that wants to test different ways to get atropine into the body). The Sponsor is the Biomedical Advanced Research and Development Authority (BARDA). BARDA is part of the United States (U.S.) Government Department of Health and Human Services. Part of BARDA's mission is to find antidotes to poisonings from chemicals and overdoses of drugs. They try to find drugs that people take regularly and ask, "Could this drug also be used to treat a poisoning?" Atropine is one such drug, it can be used to treat poisoning with a chemical called a Nerve Agent.

# 2. PURPOSE OF THE STUDY

The drug you will receive in this study is called atropine sulfate – it is an approved, marketed drug that can be given as an antidote for nerve agent poisoning of our troops or people who are exposed to these chemicals. Atropine has been approved since the 2<sup>nd</sup> World War for the treatment of nerve agent poisoning. It is most effective when given early after poisoning.

This study will help us determine if we can use another form of atropine (eye drops) to save people who have been exposed to nerve agents when the injectable form of atropine may not be readily available.

The study drug (atropine sulfate eye drops) is an approved, marketed drug often used by your eye doctor to dilate the pupils to allow for adequate examination of the back of your eye and retina.

Atropine eye drops have been given for many years off-label (outside of its approved label instruction) under the tongue ("sublingually") to manage excessive "drooling" caused by some other conditions. No serious side effects were noted with the sublingual delivery of atropine in one of the previous research studies performed before the current study.

This research study is not intended to treat any current medical condition. However, as an alternative to administration of IM atropine, atropine sulfate eye drops may be an additional source of atropine to treat chemical toxicity in an emergency setting. This bioequivalence — bioavailability and pharmacokinetics (PK) study is designed to compare how much atropine sulfate from eye drops delivered under the tongue and atropine sulfate injected into the muscle of the leg appears in the body's bloodstream. Frequent blood measurements will also allow us to determine if these different dosing routes behave similarly in the body by evaluating how the body processes the study drug.

If you qualify for the study, you will receive one dose ( $100 \,\mu\text{L}$ ) of atropine sulfate 1% eye drops sublingually (delivered under the tongue) and one dose of atropine sulfate 2.5 mL injected into thigh muscle each at 2 separate study visits. The order in which you receive these forms of the study drug will be assigned by chance, like the flip of a coin. Administration of the study drug is described below:

- A small amount of atropine sulfate 1% (2 drops or 1/10<sup>th</sup> of an mL) eye drops will be dropped under the tongue at one visit (Visit 1 or Visit 2). This is the same amount of liquid as two drops of water.
- A small amount of atropine sulfate (approximately half a teaspoon) will be injected from a syringe using a needle into the middle area of the front and side region of the thigh muscle at another visit (Visit 1 or Visit 2).

# 3. HOW LONG THE STUDY WILL LAST AND HOW MANY PEOPLE WILL BE IN THE STUDY

The study will last for 15 days and will require 3 one-day visits to the clinic. About 46 healthy men and non-pregnant women, aged 18 through 65 years, are expected to be in this study.

#### 4. TO BE IN THIS STUDY

While participating in this research study, you will need to:

- Be willing and able to a) sign this form, b) follow the study directions, and c) complete all the procedures as scheduled.
- Be in good health without certain disease conditions as specified and confirmed by the study doctor based on the check of your medical history and the results of the tests performed at the Screening Visit.
- Tell the study staff about any side effects or problems that you may face during the study.
- Ask questions as you think of them.
- Tell the study doctor or study staff if you change your mind about staying in the study.

You cannot be in this study if you:

- Are in another research study or if you have been in any other research study in the last 30 days.
- Are a woman who is pregnant or breastfeeding.
- Have taken any prescription medications (with the exception of oral contraceptives or hormone replacement therapy) within 30 days of the Screening Visit or any over-thecounter medications/vitamins/herbal supplements within 72 hours prior to the Screening Visit. Before giving each dose of study drug, the study doctor will review all the medications taken by you and decide if you can continue with the dosing or have to be discontinued from the study treatment.
- Are a smoker or use any nicotine or tobacco products such as vaping, chewing tobacco, or nicotine-containing gum, or have used any of them within 6 months before Screening.
- Plan to donate blood during the study or have donated blood within 8 weeks before Screening.
- Have a history of consuming larger amounts of alcohol or any controlled substances in the last 2 years or a positive result for urine drug test at the Screening Visit.

- Are allergic or have had any side effects to atropine in the past.
- Have consumed alcohol within 24 hours before the visits at which study drug will be given (Visit 1 and Visit 2).
- Have any condition that the study doctor may believe might put your health at risk if you participate in this study, would interfere with the routes the study drug will be given, or would interfere with the calculation of study results.

We ask that you be honest with the study doctor about your health history, or you may potentially harm yourself by taking part in this study. It is extremely important for your health and safety to tell the truth about your medical history, particularly any cardiac history, and all medications that you are currently taking or have taken within the time required for the study. For your continued safety, if you develop any new conditions or start any new medications during the study, you must inform the study doctor right away.

# Participant Responsibilities:

You will be served meals and snacks at determined times during the visits that you will receive a dose of atropine (Visit 1 and Visit 2). Please do not bring outside food or beverages, particularly caffeinated products that may interfere with study results. Some of the requirements and restrictions for this study are listed below:

- You must agree to follow all the study restrictions and rules and regulations set by the research center.
- You will be given a copy of the rules and regulations to read and sign during the Screening Visit.
- You will have to wear an identity bracelet for all the in-clinic visits (Screening, Visit 1, and Visit 2) for the entire duration that you remain in the clinic on those visit days.
- Failure to obey the restrictions, rules, and regulations of the study may lead to an end of your participation in this study which will require you to leave the study site and a possible reduction of your payment.
- You will be tested for recreational drugs or alcohol use at any time during the study per the judgement of the study doctor. If you are taken out of the study for having positive test results for drug or alcohol use, for refusing to give a specimen or providing urine samples that do not meet the temperature requirements, you will not be paid for any additional participation in this study.
  - The results of all testing in this study are confidential and never shared with anyone but study staff – in other words a positive test for recreational drugs will not be shared with law enforcement, an employer, or a family member.

#### 5. WHAT WILL HAPPEN DURING THE STUDY?

# **Screening**:

Before the study starts, you will be asked to read and sign this consent form. The study staff will thoroughly check if you are eligible to be a part of this study. Be honest while providing the details of your health history (for example, telling the study staff if you take any over-the-counter or prescription medicines, supplements, vitamins, minerals, or herbal products). You will also be asked if you currently or have ever used tobacco or vaping products and if you do use them, how often and how much.

The study doctor will conduct the tests described below to find out if you can be in the study:

- Physical examination, including height and weight
- Vital signs (temperature [by mouth], heart rate, breathing rate, and blood pressure)
- Electrocardiogram (ECG) to check heartbeat pattern: To perform the ECG, you will have stickers placed on selected locations on your chest, arms, and legs. The machine connects to these stickers and records the activity of your heart. If there is hair where the stickers need to be placed, small areas may need to be shaved. After the ECG is complete, these stickers will be removed. All the ECGs collected during the study will be checked by a medical professional for any abnormalities.
- Blood collections to check human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HbsAg), and hepatitis C antibody (anti-HCV) tests, laboratory tests, and pregnancy test for female participants. These tests will require drawing 4 or 5 tubes of blood, which amounts to less than 2-3 ounces (about 4 to 5 tablespoons [tbsp]).
  - Note: To avoid multiple needle sticks, participants will ideally have blood draw assessments done from an IV, you will be assessed for any history of prior difficulties in obtaining IV access.
- Urine sample will be collected to check for the presence of recreational drugs (e.g., amphetamines, cocaine, tetrahydrocannabinol, methylenedioxymethamphetamine, and opiates). Any positive results for recreational drug tests will be kept confidential and will not be transmitted to law enforcement authorities, unless required by a court of law.

The study doctor may determine that you are not suitable for the study based on the study plan requirements or other concerns. If you do qualify to take part in this study and you go on to participate and receive the study drug, then the following will apply:

# **Visit 1 (Day 1)**:

After completing the Screening Visit, you will be asked to return to the research site sometime within the next 3 to 14 days for Visit 1. The study staff will check if you meet the requirements to receive atropine.

You will be assigned by chance to the order in which you will receive each of the 2 different doses of atropine at your two dosing visits at the site. The order of getting the study drug is shown in Figure 5-1. You have an equal chance of being assigned to either of the 2 dosing

sequences. This is an open-label study, meaning that the study doctor, study staff, BARDA, and you will know the study drugs and the doses given to you.

Figure 5-1 Overall Study Design



There is a "washout" period between the two study treatment visits. This is designed to allow your body to remove all of the study drug from the first dose before getting the next dose. The washout period is about  $6 \pm 1$  days long.

During Visit 1, the following procedures will occur in the order mentioned below:

## Prior to study drug administration

When you return to the clinic for Visit 1 to receive study drug, you will be admitted to the research unit, you will be issued a study identification bracelet with your participant identification number, and the following will be obtained:

- Weight
- Concomitant medications (any prescription or over-the-counter medicines, vitamins, or herbal preparations) you might have taken since the Screening Visit
- Physical examination based on any symptoms you report to the study doctor or study team
- Vital signs and ECG
- Urine collection to test for pregnancy in women
- Blood collections for PK assessments
- Assessment of adverse events (AEs)/side effects
- Any alcohol, caffeine, or recreational substance use (to include nicotine and tobacco products)

You should not eat or drink anything and avoid taking any other products by mouth (even candy, chewing gum, mints, etc.) for 2 hours before you receive an atropine dose (and at least 1 hour before you arrive at the facility).

# **During study drug administration**

After fasting for a minimum of 2 hours, you will receive either atropine sulfate drops under your tongue by a pipette (a device kind of like an elaborate eye dropper that accurately measures small amounts of liquids) or atropine sulfate via injection into the middle area of the front and side region of your thigh muscle. Which of these atropine doses you receive at Visit 1 will be based on the dosing sequence determined by chance prior to you receiving the first dose. You will be asked to swallow once before you receive atropine under the tongue if that is the dose you are given that day. This is done to make sure your mouth is ready to receive the small amount of liquid that needs to be absorbed from under your tongue and to allow you to hold the study drug under your tongue for as long as possible. After receiving the study drug under your tongue, you will be informed not to swallow for at least 30 seconds. After that time, you may swallow as normal.

## After study drug administration

The following information will be collected, and the procedures and examinations listed below will be performed:

- Blood pressure and heart rate will be measured automatically every  $15 \pm 5$  minutes for the first hour, every  $20 \pm 5$  minutes for the second hour, and every  $30 \pm 5$  minutes for the third and fourth hours and thereafter as required. The readings will generally be taken on the opposite arm from which the blood has been collected.
- Blood sample collection for PK assessments will be taken at 5, 10, 15, 20, 30, 45, 60, and 90 minutes, and 2, 2.5, 4, 6, and 8 hours post dose from an IV in your arm
- ECG will be performed if the study doctor feels it is necessary or if you report any complaints like chest discomfort, lightheadedness, and/or palpitations, and repeated as needed
- Assessment of AEs and concomitant medications

You will be asked not to eat or drink for 2 hours after an atropine dose has been given or until you start experiencing unbearable dryness in your mouth. You will be offered water as needed after 2 hours or as you complain of intolerable dryness in mouth. You will be given a meal/snack approximately 4 hours after study drug administration. You will be released from the clinic after the 8-hour post-dose blood sample collection.

#### Visit 2 (Day $8 \pm 1$ day):

After Visit 1, you will need to return to the clinic in about 7 days for Visit 2. This gap of 6  $(\pm 1)$  days in between is called as washout period, and it is necessary to allow your body to be completely free of the previous dose of atropine. Visit 2 will be like Visit 1 with respect to dosing and procedures, except that you will receive the other type of atropine dose that you did not receive at Visit 1.

# Telephone Follow-up Visit (Day 15 -1/+7 days)

At the conclusion of your time in the study, you will have a follow-up telephone call from the clinic about 7 days after you leave the clinic following your Visit 2. During this call, you will be asked if there were any changes in your general health and if you have taken any medications (over-the-counter or prescription medicines, vitamins, minerals, or herbal products) AFTER you left the clinic following your second dose. The purpose of this call is to gather information on any changes to your health.

#### 6. BLOOD SAMPLES COLLECTED DURING THE STUDY

Blood samples for checking eligibility at Screening will be taken from either your left or right arm using a needle and a collection vial. About 8 teaspoons (40 mL) of blood will be drawn at the Screening Visit.

A total of two teaspoons (10 mL) of blood will be collected at each blood draw time point. This blood will be used to determine how your body is processing the atropine dose at Visits 1 and 2. If the IV cannot be used at any time point, it may be necessary for the blood sample to be drawn using a needle stick (normal way a blood test is collected) if there is no alternative. You may not be able to choose how a blood sample is obtained, but refusing a sample collection may require you to opt out of the study at that point. There will be 14 blood draws in each single dosing visit for PK samples. Since a catheter will be used to collect the PK blood samples, a small amount of blood will be drawn and discarded to clear the line before each PK blood draw. The amount of blood drawn to be discarded is approximately 84 mL (about 1/3 cup). The total amount of blood drawn over the study will be less than 280 mL (1.25 cups). For comparison, the standard blood donation is about 480 mL (2 cups).

#### 7. HIV AND HEPATITIS TESTING

As required by the study, you must have your blood tested for the HIV and hepatitis viruses. HIV is the virus that causes acquired immunodeficiency syndrome (AIDS). If you have a positive HIV or hepatitis test result, you cannot participate or continue in the study.

If the HIV test is positive, a follow-up test will be done. If the follow-up test also shows a positive result, you will be told about it in private and will be given counselling.

In the interest of public and participant safety, if we cannot reach you by phone to provide you with the HIV, Hepatitis B and/or Hepatitis C results, or you do not respond to the return receipt letter, we will send the positive results to your address available in our records via a certified mail.

It may take 2-3 months after being infected with HIV for the test to be positive. The HIV test does not always give correct results.

Positive test results are required to be reported to the State Department of Health. If you have any questions about what information is required to be reported, please ask the study doctor or any other staff member.

Although this testing is supposed to be private, this cannot be guaranteed. For example, it is possible for a court of law to get health or study records without your permission as per Health Insurance Portability and Accountability Act compliance, individual authorization as required at 45 Code of Federal Regulations (CFR) 164.508 or with a waiver of individual authorization as permitted at 45 CFR 164.512(i).

#### 8. POSSIBLE SIDE EFFECTS AND RISKS OF ATROPINE SULFATE

You must tell the study doctor or study staff about all side effects that you may experience during the study. If you are not honest about your side effects, you may harm yourself by continuing in this study.

There may be risks associated with atropine that are not currently known; however, below is a list of the most common side effects of atropine sulfate ophthalmic solution, USP 1%, when administered in the eye(s):

- Sensitivity to light
- Blurred vision
- Eye pain/stinging
- Reduced tears
- Dry skin, mouth, and throat
- Increased blood pressure
- Increased heart rate, heart may feel like it is beating fast
- Restlessness
- Irritability/confusion
- Flushed skin
- Allergic reactions

As reported in many published medical articles, atropine sulfate ophthalmic solution has been given safely to over 400 people under the tongue. The most common side effect has been dry mouth.

Below is a list of the most common side effects of atropine sulfate injection solution given via IM injection:

• Increased heart rate (with recurrent use)

- Increased blood pressure
- Dry skin, mouth, and throat
- Blurred vision
- Increased eye pressure
- Intestinal problems like constipation and in rare cases a blockage
- Trouble urinating
- Thickening of mucus
- Flushed skin
- Trouble with producing sweat
- Headache
- Confusion
- Dizziness
- Nausea or vomiting
- Fatigue (tiredness)

These effects are generally short-lived and go away within hours. You will be monitored closely for any of these symptoms after you have received atropine at each visit.

Administration of the study drug, like any drug, may cause an allergic reaction. You will be monitored carefully after administration of the study drug for signs of an allergic reaction. There are trained medical staff, emergency equipment and medicines available at the study site to treat you in the event of an allergic reaction. Symptoms of any allergic reaction can include a rash, hives, itching, and/or difficulty in breathing, closing of the throat, and swelling of the lips, tongue, or face. It may rarely cause death. If you experience any of the above symptoms or any other significant symptoms after you leave the clinic, dial 9-1-1 and seek medical attention immediately, and notify the study staff listed on the first page of this consent document.

Participants who develop any visible skin reaction may have the area photographed to document the extent of the reaction. These photographs will only be labeled with your participant ID number and will not contain any personal information.

Until you know how the study drug will affect you, you should use caution by avoiding stairs, not driving a car, and not working with machinery. However, the side effects, if any, of this study drug is generally short-lived and is not anticipated to persist longer than your scheduled visits. However, you may want to consider having someone driving you to the clinic and picking you up if you are sensitive to medicines.

If you do not understand what any of these side effects mean, please ask the study doctor or study staff to explain these terms to you.

# 9. ADDITIONAL RISKS OR DISCOMFORTS

#### Blood collection:

There are some side effects of collecting blood at the Screening Visit and for PK samples at Visits 1 and 2.

Possible side effects of collecting blood include:

- Fainting
- Redness
- Pain
- Bruising
- Bleeding
- Infection
- Nerve damage
- Blood clots, which may cause inflammation, swelling and pain

If you feel you are about to pass out, tell the study staff immediately.

# Electrocardiogram:

The ECG test is a recording of the electrical activity of your heart. The sticky pads used may be cold when applied and sometimes cause some discomfort such as redness or itching. If the hair under the patches needs to be shaved, irritation from shaving could occur. Sometimes hair may be removed when the sticky pads are removed. All efforts will be made to avoid this inconvenience.

# Risks of IM injection:

- Pain
- Redness
- Bruising
- Irritation from the fluids or drug being given
- Local swelling
- Accidental injecting into the underlying nerves, blood vessels, or bone (if the needle of the injection is too long)
- Infection is a serious, but very rare risk
- Fainting

# 10. BIRTH CONTROL, DANGERS OF PREGNANCY AND BREAST FEEDING

If you are a female, you should avoid the possibility of becoming pregnant while in this study. The only certain way to not get pregnant is to not have sex. If you are a female of childbearing potential (able to become pregnant) and choose to have sex with a male partner, you must use one of the following methods of birth control for at least 2 months before the Screening Visit and agree to continue using an acceptable form for the duration of the study (from the Screening Visit through Follow-up Visit [Day 15]).

Adequate contraception is defined as a contraceptive method with a failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label. Some of the examples of contraceptive medications include:

- Oral contraceptives
- Injectable progestogen
- Implants of etonogestrel or levonorgestrel
- Estrogenic vaginal ring
- Percutaneous contraceptive patches
- Intrauterine device (IUD) or intrauterine system
- Male partner sterilization at least 6 months prior to the female participant's Screening Visit

A female of childbearing potential is defined as a post onset of menarche and premenopausal female capable of becoming pregnant. This does not include females who meet any of the following conditions:

- Menopausal greater than 2 years
- Tubal ligation (tubes tied) greater than 1 year
- Bilateral salpingo-oophorectomy (removal of both ovaries and fallopian tubes)
- Hysterectomy (removal of the uterus)

Even if you use birth control during the study, if you are female, there is still a chance you could become pregnant. If you are pregnant or become pregnant during the study, the study drug may pose unexpected risks to the unborn baby. A pregnancy test does not always show correct results, especially in the early stages of pregnancy.

If you become pregnant from the start of Visit 1 until the Telephone Follow-up Visit is finished, inform the study doctor or study staff member immediately. You will not be given any further doses of the study drug once your pregnancy gets confirmed. The study doctor will counsel you on the harmful effects of continuing in the study and the possible effects of the study drug on the baby. You will be closely observed until you deliver the baby. If you have an abortion (suggested

by the doctor), miscarriage, or notice birth defects in the baby, please let the study staff know about it right away.

Similarly, you cannot be in the study if you are breastfeeding. It is not known whether the study drug can be given to mothers who breastfeed their babies. Therefore, if you are breastfeeding a child, you cannot participate in this study.

#### 11. POSSIBLE BENEFITS OF PARTICIPATING IN THIS STUDY

This study is for research purposes only. You will get no medical benefit from this study. Information learned from this study may help other people in the future.

# 12. ALTERNATIVES TO PARTICIPATING IN THE STUDY

As this study is for research purpose only, the only other choice would be not to take part in the study.

#### 13. CONFIDENTIALITY

This research is covered by a Certificate of Confidentiality (CoC) from BARDA, Administration for Strategic Preparedness and Response, a US Federal Government entity under Health and Human Services.

This means that the staff of BARDA, Rho, Inc., Allucent, Johnson County Clin-Trials (JCCT), and Institutional Review Board (IRB, the committee which reviews the study as related to safety and risk-benefits) cannot share or give to any other person not connected with this research your name, information about you, documents, or samples that may identify you in any action or suit unless you say it is okay.

A CoC protects your private information from all legal proceedings. Your information cannot be used as evidence even if there is a court subpoena. All copies of your information are immune from the legal process, and cannot, be admitted as evidence or used for any purpose in any action, suit, or other judicial, legislative, or administrative proceeding unless you say it is okay.

The information about you CAN be shared for other research if it is allowed by federal regulations. We will let you know beforehand if this is something we will do.

The Certificate DOES NOT stop the reporting that federal, state, or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop the U.S. federal or state government agency from checking records or evaluating programs. The Certificate DOES NOT stop disclosures required by the federal Food and Drug Administration (FDA).

You should understand that a CoC does not keep you from voluntarily releasing information about yourself or your involvement in this research. It also does not prevent you from having access to your own information. If you want your research information released to an insurer,

medical care provider, or any other person not connected with the research, you must provide specific consent to allow the researchers to release it.

Your information or the biological samples (blood samples collected to measure atropine levels) will not be used or distributed for future research studies even if identifiers have been removed.

Your biospecimens collected during this study may be used for commercial profit (even if identifiers are removed) and you will not share in this profit.

Research results that are clinically relevant, including individual research results, will not be disclosed to you.

Researchers can look closely at large amounts of your genetic information by sequencing, or "reading," every letter in your DNA (your genome). Reading a person's entire genetic code is called whole genome sequencing. The research will not include whole genome sequencing (for example, sequencing of a human germline or somatic specimen with the intent to generate the genome or exome sequence of that specimen).

A description of this clinical trial will be available on <a href="www.ClinicalTrials.gov">www.ClinicalTrials.gov</a>, as required by the U.S. Law. This Web site will not include information that could identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

The IRB, the FDA, and accrediting agencies may inspect and copy your records, which may have your name on them. Therefore, total confidentiality cannot be guaranteed. If the study results are presented at meetings or printed in publications, your name will not be used.

#### 14. IN CASE OF STUDY RELATED INJURY

If you become ill or are injured while you are in this study, ask for medical care right away and notify the study staff listed on the first page of this consent form. You should inform the healthcare professional treating you about your participation in this study.

The study doctor may ask you to stay longer at your current visit, have additional testing or return to the clinic for an additional visit. If you tell the study staff that you think you have been injured, the study staff may ask you to visit the clinic or refer you to other medical care providers for medical care, even after you have completed your regular study visits.

If you are injured as a result of taking the study drugs or from procedures done for the purpose of this study, Allucent will pay for those medical expenses necessary to treat your injury that are not covered by your medical insurance or any other third-party coverage. You will not lose any of your legal rights or release BARDA, the study doctor, the study staff, or study site from legal responsibility for mistakes by signing this consent document.

To pay medical expenses, Allucent will need to know some information about you like your name, date of birth, and Medicare Beneficiary Identifier (MBI). This is because Allucent must check whether you receive Medicare and, if you do, report the payment it makes to Medicare.

The study drug and the clinical trial are covered by the Public Readiness and Emergency Preparedness (PREP) Act which limits your ability to sue if you develop a reaction to the study drug. A federal program has been created to help pay for medical care and other specific expenses of people who have serious reactions that are caused by the study product. To be eligible for this program, you must file a claim within one year of receiving the study drug. The program is administrated by the Health Resources and Services Administration. An information sheet about the PREP Act and the Federal program, including how to file a claim, will be provided to you http://www.hrsa.gov/cicp/.

#### 15. LEGAL RIGHTS

You will not lose any of your legal rights by signing this consent form.

#### 16. WHOM TO CONTACT ABOUT THIS STUDY

During the study, if you experience any medical problems, suffer a research-related injury, or have questions, concerns or complaints about the study such as:

- Whom to contact in the case of a research-related injury or illness;
- Payment or compensation for being in the study, if any;
- Your responsibilities as a research participant;
- Eligibility to participate in the study;
- The study doctor's or study site's decision to withdraw you from participation;
- Results of tests and/or procedures.

# <u>Please contact the study doctor at the telephone number listed on the first page of this consent document.</u>

If you seek emergency care, or hospitalization is required, alert the treating physician that you are participating in this research study.

An institutional review board (IRB) is an independent committee established to help protect the rights of research participants. If you have any questions about your rights as a research participant, contact:



Please reference the following number when contacting the

### 17. COSTS

There will be no charge to you for your participation in this study. The study drug, study-related procedures, and study visits will be provided at no charge to you or your insurance company

#### 18. PAYMENT FOR BEING IN THIS STUDY

You may receive up to \$ for taking part in this study. You will be paid per completed visit as follows:

| Visits | Compensation (amount in \$) |
|--------------------------|-----------------------------|
| Screening | |
| Visit 1 | |
| Visit 2 | |
| Follow-up Telephone Call | |

Total compensation will be up to \$ for completion of all study visits and the follow-up telephone call. If it is determined by your study doctor that you should stop the study early, or you choose to withdraw from the research study, the payment will be prorated based on the study visits you complete as detailed in the table above. This means you will only be paid for the study days you participate in. If you check-in to the facility for Visit 1 or Visit 2 and get discharged from the study prior to that day's dosing and thus not completing that day's scheduled activities, you will receive \$ as compensation within seven (7) days of study completion.

The amount provided for each visit is intended to provide you with financial support for travel and the cost of inconvenience for participating in this clinical study. Please ensure you bring enough funds with you for transport back home from the clinic for all visits. You will receive your compensation within seven (7) days of study completion.

If it is necessary for JCCT to obtain medications, study supplies that you were supposed to provide, clothing, toiletries, or transportation outside of what is described in this consent, you will be responsible for these costs. If you are unable to pay the fees upfront, JCCT will pay for these expenses and may deduct the cost from your stipend check. JCCT is not liable for your safety during travel to and from our site.

If it is necessary for you to return to the research unit for additional safety follow-up visits, you will be compensated for a completed unscheduled visit at JCCT. For more information, please talk to your study doctor.

No deductions will be withheld from your compensation check for tax purposes. You will be responsible for reporting any payment on your state and federal tax returns. Your involvement in this study does not make you an employee of BARDA or the study site. At the end of each year, the study site will notify the Internal Revenue Service of all stipends you have received

throughout the year. If the compensation you received is over \$ 900, you will be issued a 1099 form by JCCT.

#### 19. VOLUNTEERING TO BE IN THE STUDY

It is completely your choice to be in this study, and no one can force you to be a part of this study. If you do not want to continue in the study, you may leave at any time without penalty or loss of any legal rights to which you are otherwise entitled.

If you meet one or more of the conditions stated below, you will be kept off of the study drug for some period of time until the study doctor discusses with the medical monitor and BARDA about the scenario.

- You experience any severe or higher-intensity AE that in the opinion of the study doctor is possibly caused by the study drug.
- You experience an AE that might require a treatment, observation for safety, or limits some of the body functions, thereby making further dose administration inappropriate.
- You no longer meet eligibility criteria, and it is not safe for you to continue in the study.

You will be recommended to either continue to receive study drug per the study plan or discontinue further dosing once your condition has been reviewed by the medical monitor and BARDA.

The study will be kept on hold for all participants, if:

- Two or more participants experience a severe reaction in the same part of the body and the medical research staff consider the reactions as possibly related to the study drug.
- One death possibly related to the study drug has been reported.

The study doctor, BARDA, or the FDA may take you out of the study without your permission, at any time, for the following reasons:

- If you do not follow the study doctor's instructions
- If we find out that you should not be in the study
- If the study is stopped
- If it becomes harmful to your health
- If you become pregnant
- At the request of BARDA
- At the request of IRB

If information generated from this study is published or presented, your identity will not be revealed. If you choose to leave the study by yourself or if you are taken out of the study for some reason before Day 15, you may be asked to return to clinic for a final visit to have some end of study evaluations or tests. If you leave the study early, an Early Termination (ET) visit

will be performed, when possible. The ET visit may be conducted in the clinic or by phone as determined by the study doctor. If the study doctor determines that the ET visit should be conducted in the clinic, then a physical examination (based on your symptoms) including weight, vital signs, ECG, blood samples for laboratory tests, urine sample to check pregnancy, and assessment of AEs/side effects and concomitant medications will be performed at study doctor's discretion.

#### 20. NEW FINDINGS

If there is new information or any important new findings that could relate to your willingness to continue participation, we will tell you. You can then decide if you still want to be in the study.

# 21. AGREEMENT TO BE IN THE STUDY

Please answer **YES** or **NO** to the following questions:

If you do not feel that you will be able to comply with any of the restrictions or procedures, please discuss with the study staff prior to signing and dating this consent form.

This consent form contains important information to help you decide if you want to be in the study. If you have any questions that are not answered in this consent form, ask one of the study staff members.

| | | <i>U</i> 1 |
|---|---|---|
| A. | Is this document i | this document in a language you understand? |
| | □ Yes | $\square$ No |
| В. | Has the study doc the study? | as the study doctor clearly explained the nature, benefits, and risks of your participation in the study? |
| | □ Yes | $\square$ No |
| C. | Do you understan | Oo you understand the information in this consent form? |
| | □ Yes | $\square$ No |
| D. | Have you been given enough time to ask questions and talk about the study? | |
| | □ Yes | $\square$ No |
| E. | Have all your questions been answered to your satisfaction? | |
| | □ Yes | $\square$ No |
| F. | Do you think you received enough information about the study? | |
| | □ Yes | $\square$ No |
| G. | 6. Do you volunteer to be in this study of your own free will and without feeling pressured the study doctor or study staff? | |
| | □ Yes | $\square$ No |
| H. Do you know that you can leave the study at any time without giving a reason and w your decision affecting your health care in any way? | | |
| | □ Yes | $\square$ No |
| I. | Do you know that your health records from this study may be reviewed by BARDA scientists involved in performing this study? | |
| | □ Yes | $\square$ No |

| _ <b>\</b> | Yes [ | 0 | |
|---|---|---|---|
| | you permit<br>atropine adı | be contacted with a request to participate in future clinical saistration? | tudies related |
| to a | - | cipating in this clinical trial, the sponsor may have future opport stration, your selection below does not impact your ability to par | |
| | □ Yes | □ <b>No</b> | 1 |
| L. | L. Are you aware that you will not be refused care at the JCCT, where the staff are trained in ACLS and other lifesaving care to stabilize your condition before you reach the hospital. | | |
| | □ Yes | $\square$ No | |
| K. | . Are you aware that Johnson County Clin-Trials (JCCT [Address: 16400 College Blvd, Lenexa, KS 66219, United States]), is a research facility and not a place for routine medical care but is the first place to report any study-related complaint. Therefore, you should continue to obtain your routine medical care with the provider of your choice. Are you also aware that JCCT will refer you to outside medical care if treatment is needed as a result of the study drug or study procedures. | | |
| | □ Yes | $\square$ No | |
| J. | Do you kno | hat you cannot be in another clinical trial or study while you are | in this study? |

# IF YOU ANSWERED "NO" TO ANY OF THE ABOVE QUESTIONS, OR YOU ARE UNABLE TO ANSWER ANY OF THE ABOVE QUESTIONS, YOU SHOULD NOT SIGN AND DATE THIS CONSENT FORM

| Printed Name of Adult Participant | Time |
|-------------------------------------------|------|
| Signature of Adult Participant | Date |
| Printed Name of Person Explaining Consent | Time |
| Signature of Person Explaining Consent | Date |

You will be given a signed and dated copy of this consent form to keep it for yourself.

# 22. AUTHORIZATION TO USE AND DISCLOSE PROTECTED HEALTH INFORMATION

If you decide to be in this study, the study doctor and research team will use and share health data about you to conduct the study. Health data may include:

- Your name
- Year of birth
- Medical history
- Information from your study visits, including all test results, as described in the previous sections.

Health data may come from your study records or from existing records kept by your doctor or other health care workers.

All reasonable efforts will be taken to keep all medical records and research materials confidential. All data which are collected and obtained for the purpose of the study will only be stored, evaluated, and possibly forwarded in a coded form. Coded means that neither your name nor initials will be documented, only a number and/or a letter code, possibly together with your year of birth. The code which is required to match the coded data with your name is accessible only to the study doctor and his/her study staff, monitors, and auditors, as required. If the results of this study are published in the medical literature, you will not be identified by name.

For this study, the research team may share coded health data about you with authorized users. Authorized users generally are:

- Representatives of BARDA, the Sponsor.
- Representatives of JCCT, the research center.
- Representatives of Allucent, a Contract Research Organization that is coordinating and monitoring the study.
- Representatives of Rho, Inc, a Contract Research Organization that is coordinating the study.
- Representatives of IRB (an Institutional Review Board that reviews this study, safety, and ethics and to ensure participant's rights are not violated).
- The FDA and other U.S. federal and state agencies for the purpose of ensuring that the medical information was collected ethically and accurately.
- Government agencies to whom certain diseases (like HIV, hepatitis, and sexually transmitted diseases) must be reported in response to lawful requests and law enforcement requirements.
- Outside individuals and companies, such as laboratories and data storage companies, that work with the researchers and BARDA and need to access your information to conduct this study, store data or analyzing study results.

• A data safety monitoring board which oversees this research, if applicable.

Your health data will be used to conduct and oversee the research, including for instance:

• Other research activities related to the study drug.

Once your coded health data has been shared with authorized users, it may no longer be protected by federal privacy law and could possibly be used or disclosed in ways other than those listed here.

The monitors, the auditors, the IRB, and the regulatory authority(ies) will be granted direct access to your original medical records for verification of clinical trial procedures and/or data, without violating your confidentiality, to the extent permitted by the applicable laws and regulations. By signing this form, you are authorizing such access.

Your address and telephone number may be collected by the study doctor for the purpose of the Institution's legal requirement of submitting taxes to the IRS. This data will not be used for the study, nor stored in any study files or shared with BARDA or its representatives.

The research team's permission to use and share health data about you will end in 50 years unless you revoke it (take it back) sooner.

You may revoke (take back) your permission to use and share health data about you at any time by writing to the study doctor. If you do this, you will not be able to stay in this study. No new health data that identifies you will be gathered after your written request is received. However, health data about you that has already been gathered may still be used and given to others as described in this form.

Your right to access your health data in the study records will be suspended during the study to keep from changing the study results. When the study is over, you can access your study health data.

If you decide not to sign and date this form, you will not be able to take part in the study.

# 23. STATEMENT OF AUTHORIZATION

| I have read this form, and its contents were explained to me clearly. My questions have been answered. I voluntarily agree to allow study staff to collect, use and share my health data as specified in this form. I will receive a signed and dated copy of this form for my records. I am not giving up any of my legal rights by signing and dating this form. | |
|---|---|
| □ I <b>Voluntarily Agree</b> to allow study staff to collect, use and share my health data as specified in this form. | |
| □ I <b>DO NOT Agree</b> to allow study staff to collect, use and this form, therefore, I am unable to participate in the study. | share my health data as specified in |
| Printed Name of Participant | |
| Signature of Participant | Date |
| Printed Name of the Person Obtaining the Authorization | |
| Signature of the Person Obtaining the Authorization | Date |